CLINICAL TRIAL: NCT00005499
Title: Congestive Heart Failure Trends in the Elderly 1970-94
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5017; R01HL058880 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2004-08

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Heart Failure, Congestive; Heart Failure
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Heart Failure

SUMMARY:
To investigate trends in the incidence and survival rates of congestive heart failure (CHF) in two successive cohorts of elderly people (1970-74, 1990-94) in a health maintenance organization (HMO).

DETAILED DESCRIPTION:
BACKGROUND:

The study constituted part of a growing body of research designed to understand not only the secular trends in mortality, morbidity, survival, and disability levels for selected major chronic diseases among older persons in the United States, but also the implications of the findings for health care utilization.

DESIGN NARRATIVE:

The design was that of a retrospective study of successive cohorts of a well-defined and well-documented elderly population for the purpose of identifying and explaining trends in congestive heart failure (CHF) incidence, survival, comorbidities and health services utilization during the 25-year period 1970-1994. The study sample consisted of two successive period cohorts of elderly people, identified for each of two five-year periods, 1970-1974 and 1990-94. The study tested the following hypotheses: 1) incidence of CHF had decreased among the younger old (65-74 years of age); 2) incidence of CHF had increased among the older old (75 years of age or above); 3) one-year survival time had increased following onset of incident CHF; and 4) prevalence of hypertension had decreased and prevalence of myocardial infarction and other manifestations of coronary artery disease increased among incident cases of CHF.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-07; Study Completion 2001-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Barker — Kaiser Foundation Research Institute